CLINICAL TRIAL: NCT01023776
Title: Evaluation of the Infectivity, Replication, and Immunogenicity of Live, Attenuated A/California/07/09 (nH1N1) Influenza Vaccine in Serosusceptible Adults
Brief Title: Infectivity, Replication & Immunogenicity of Live nH1N1 Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, John Treanor, M.D., University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: URMC 09-006
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-11

CONDITIONS: Influenza
Keywords: Swine Flu; H1N1
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- live monovalent H1N1 vaccine (Other): A/California/07/09 live monovalent H1N1 vaccine 0.2 given intranasally, 2 doses given 28 days apart
  Interventions: Biological: A/California/07/09 live monovalent H1N1 vaccine

INTERVENTIONS:
Biological: A/California/07/09 live monovalent H1N1 vaccine — 0.1mL per nares intranasally, second identical dose given 28 days after first vaccine
  Other Names: Influenza A (H1N1) 2009 Monovalent Vaccine Live, Intranasal

SUMMARY:
The purpose of the study is to determine the amount of live virus that can be recovered from the nose of people who are vaccinated with the licensed live vaccine against H1N1, and to describe the immune response to vaccination.

DETAILED DESCRIPTION:
By looking at the immune response before and after vaccine, we hope to understand the factors that determine the immune response and detailed shedding patterns of live novel H1N1 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-32 years, inclusive
* No history of Novel H1N1 virus or vaccine
* Female not able to bear children or not pregnant and agrees to practice effective birth control
* Female negative pregnancy test
* Good Health
* Ability to understand and comply with protocol
* Provided Informed Consent

Exclusion Criteria:

* Previous history of vaccination against novel H1N1 or laboratory documented H1N1 infection
* History of egg allergy or is allergic to other components of the vaccine
* A women who is pregnant or breastfeeding or intends to get pregnant during the study period between enrollment and 30 days following vaccination
* Subject is immunosuppressed as the result of underlying illness or treatment with immunosuppressive or cytotoxic drugs or use of chemotherapy or radiation therapy in the preceding 36 months
* Subject has active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematological malignancy. "active is defined as treatment within the past 5 years
* Long term (greater than 2 weeks) use of oral or parental steroids, or high- dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids allowed)
* Received immunoglobulin or another blood product within 3 months prior to enrollment in this study
* Subject has received an inactivated vaccine within 2 weeks or a live vaccine within 4 weeks prior to enrollment in this study or plans to receive another vaccine within the next 28 days (or 56 days for the vaccine naive recipients)
* Subject has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses. Those conditions include chronic conditions recognized as risk factors for influenza complications or as contraindicated for live vaccination, including chronic cardiac (exclusive of hypertension) or pulmonary conditions (including asthma), diabetes mellitus, or renal impairment
* Subject has an acute illness or an oral temperature greater then 99.9 degrees F(37.7 C)within 3 days prior to enrollment or vaccination. Subject who has acute illness that was treated, symptoms resolved are eligible to enroll as long as treatment is complete and symptoms resolved > 3 dyas prior to enrollment.
* Subject is currently participating or plans to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication) or has received an experimental agent within 1 month prior to enrollment in this study, or intends to donate blood during this period.
* Subject has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
* Subject has a history of alcohol or drug abuse in the 5 years prior to enrollment.
* Subject has known human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Subject has a previous history of Guillain-Barre syndrome within 6 weeks of receipt of influenza vaccine
* Subject has any condition that the principal investigator (PI) believes may interfere with the successful completion of the study

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J. Treanor, M.D., Principal Investigator — University of Rochester
Locations (1):
- Vaccine Research Unit Room 3-5000, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy Volunteers were recruited from the general public between December 2009 and January 2010
Pre-assignment Details: 28 volunteers were recruited; 20 were enrolled and received at least 1 dose of vaccine, 8 were excluded (2 refused further participation and 6 did not meet inclusion criteria #2)
Groups:
- Live Monovalent H1N1 Vaccine: Subjects received 2 doses of vaccine 0.1 ml in each nostril intranasally 28 days apart
Period: Overall Study
Arm/Group | Live Monovalent H1N1 Vaccine
Started | 20 (Subjects received 2 dose of vaccine 0.1 ml in each nostril intra nasally 28 days apart)
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Live Monovalent H1N1 Vaccine: Live Monovalent H1N1 vaccine 0.1 ml in each nostril times 2 doses given intranasally 28 days apart
Arm/Group | Live Monovalent H1N1 Vaccine
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (3.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Shed Virus
Description: number of participants who shed virus above the limit of detection at any timepoint after vaccine. The limit of detection is 0.5 tissue culture infectious doses per mL of nasal wash.
Time Frame: 28 days post vaccine 1 and 28 days vaccine 2
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Live Monovalent H1N1 Vaccine
Number analyzed (Participants) | 20
participants | 0

2. Secondary Outcome: Mean Difference Between Cycle Time and Detection Threshold
Description: The mean difference was calculated by real-time polymerase chain reaction (PCR) on nasal wash samples. Cycle time is the cycle number at which the PCR reaction is positive with a range of 0-40 cycles. The detection threshold is 40 cycles.
Time Frame: day 10 post vaccine 1
Population: per protocol
Measure: Mean (95% Confidence Interval); unit: cycles
Arm/Group | Live Monovalent H1N1 Vaccine
Number analyzed (Participants) | 20
cycles | 0.0075 [.001 to .01]

ADVERSE EVENTS:
Time Frame: 56 days
Description: Participants were queried at each visit about the occurence of any adverse events.
Arm/Group | Live Monovalent H1N1 Vaccine
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 11/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Live Monovalent H1N1 Vaccine (N=20)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Light Headed (Nervous system disorders) | 1 (1)
Menstral Cramps (Reproductive system and breast disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Swollen glands (Blood and lymphatic system disorders) | 2 (2)
URI (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No